CLINICAL TRIAL: NCT05372913
Title: A Randomized Controlled Trial of the Feasibility and Acceptability of W-GenZD Versus CBT-light Teletherapy for Adolescents Seeking Mental Health Services
Brief Title: Feasibility and Acceptability of W-GenZD vs CBT-light Teletherapy for Adolescents Seeking Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Woebot Health (Industry)
Collaborators: Children's Hospital of The King's Daughters (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W-GenZD-003
Record Dates: First submitted 2022-04-29; First posted 2022-05-13 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety
Keywords: Mental Health; Adolescence; Digital Therapeutic; Cognitive Behavioral Therapy; Chatbot; Mental Health App
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-GenZD Mobile Application Group (Experimental): Participants assigned to the W-GenZD mobile application group will be asked to download and use the W-GenZD mobile application that will provide information and tools through a chatbot (a computer program designed to communicate with users). Participants will be invited to use the mobile application as often as they like during the 4-week treatment period - we will encourage 5 to 10 minutes of daily use.
  Interventions: Device: Woebot for Adolescents (W-GenZD) Mobile Application
- CBT-Lite Teletherapy Group (Active Comparator): Participants assigned to the CBT-lite teletherapy group will be asked to attend 1-hour teletherapy group sessions over Zoom once a week for 4 weeks. In this group, a study clinician will cover topics such as building a coping tool box, accepting your feelings, challenging negative thoughts, and problem solving.
  Interventions: Behavioral: CBT-Lite Teletherapy Group

INTERVENTIONS:
Device: Woebot for Adolescents (W-GenZD) Mobile Application — Woebot for Adolescents (W-GenZD) is a mobile application program that delivers evidence-based therapy for the symptoms of mild-moderate depression and anxiety in adolescents in brief "conversations" with a fully automated relational agent called Woebot. It is a brief, self-guided 4 week-intervention that draws from cognitive behavioral therapy (CBT), interpersonal psychotherapy for adolescents (IPT-A), and elements of dialectical behavior therapy (DBT), depending on the presenting situation, to help the adolescent develop emotion regulation skills in the context of their everyday life. In this way, the mobile application is designed to be targeted, relevant, and integrated into the lived experience of adolescents, capable of delivering the appropriate technique for the problem at hand, at the time of need.
  Arms: W-GenZD Mobile Application Group
Behavioral: CBT-Lite Teletherapy Group — The CBT-Lite teletherapy group is a brief, 4-week intervention held once weekly for an hour, and limited to those triaged into the Children's Hospital of the King's Daughters low-intensity track and participating in this protocol. An assigned study clinician will facilitate each teletherapy group with approximately 10 adolescents in each session. Each group begins with orientation and reviewing group rules, individual check-ins with each participant (rating stress level and hopefulness), followed by a guided mindfulness moment. Sessions are designed to draw from elements of cognitive behavioral therapy (CBT) and the 4 topics include: building a coping tool box, accepting your feelings, challenging negative thoughts, and problem solving.
  Arms: CBT-Lite Teletherapy Group

SUMMARY:
The primary aim of this study is to determine the feasibility and acceptability of the W-GenZD mobile application among a group of adolescents and who have screened and triaged into low-intensity treatment within the Children's Hospital of the King's Daughters. The secondary aim of this study is to determine the preliminary comparative efficacy of W-GenZD and CBT-light teletherapy zoom groups to manage mood concerns at 4-weeks end of treatment relative to baseline. The third aim of this study is to investigate potential differences between group differences on working alliance. An exploratory aim of this study is to observe and describe the utilization and outcomes of the safety procedures utilized within this study.

ELIGIBILITY:
Inclusion Criteria:

1. Have completed triage at the Children's Hospital of the King's Daughters (CHKD) and have been deemed appropriate for the low-intensity intervention track, given presenting problem(s) of depressive or anxiety symptoms
2. Adolescent 13-17 years of age, inclusive
3. U.S. resident
4. Both adolescent participant and parent/guardian are able to read and write in English
5. Own or have regular access to a smartphone (Android or iOS smartphone with a recent, supported operating system), that can receive SMS messages, and reliable Wi-Fi access or sufficient data to engage with assigned treatment condition for the duration of the study
6. If currently prescribed antidepressant medications (e.g. escitalopram/Lexapro, fluoxetine/ Prozac), antipsychotic medications (e.g. aripiprazole, asenapine, olanzapine, paliperidone, quetiapine, risperidone), or stimulants (e.g. amphetamine/Adderall, Methylphenidate/Ritalin) and alpha agonists (e.g. atomoxetine/Strattera, Guanfacine/Intuniv) they are at a regular, stable dose for at least 60 days at screening
7. Not currently actively engaged is psychotherapy
8. Available and committed to engage with the program and complete assessments for a 8-week duration
9. Family is willing and able to engage in discussion of safety planning in the event of suicidal symptoms

Exclusion Criteria:

1. Lifetime diagnosis of a psychotic disorder (including schizophrenia or schizoaffective disorder)
2. Lifetime diagnosis of bipolar disorder
3. Lifetime diagnosis of autism spectrum disorder or pervasive developmental disorder (e.g. autism, Asperger syndrome, Rett's syndrome)
4. Current diagnosis of developmental delay or intellectual disability
5. Suicidal ideation with a plan or intent or a suicidal attempt within the past 12 months
6. History of (a) drug and/or alcohol abuse within the past 12 months
7. Current use of benzodiazepines (e.g. lorazepam, clonazepam, alprazolam, diazepam, triazolam) or certain sleep aids (zolpidem, eszopiclone, zaleplon)
8. Previous Woebot application use
9. Enrollment of more than one member of the same household

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Margaret Gleason, MD, Principal Investigator — Children's Hospital of The King's Daughters
Locations (1):
- Children's Hospital of The King's Daughters, Norfolk, Virginia, United States

REFERENCES:
- [Derived] Gleason MM, Flom M, Rapoport S, Williams A, Birch A, Wells NK, Forman-Hoffman V, Robinson A. A Relational Agent Intervention for Adolescents Seeking Mental Health Treatment: Outcomes From a Randomized Controlled Trial Within a Children's Outpatient Hospital. JAACAP Open. 2025 Feb 11;3(4):1033-1045. doi: 10.1016/j.jaacop.2025.02.002. eCollection 2025 Dec. PMID 41367963
- [Derived] Chiauzzi E, Robinson A, Martin K, Petersen C, Wells N, Williams A, Gleason MM. A Relational Agent Intervention for Adolescents Seeking Mental Health Treatment: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 3;12:e44940. doi: 10.2196/44940. PMID 36867455

RESULTS

PARTICIPANT FLOW:
Groups:
- W-GenZD Mobile Application Group: Participants assigned to the W-GenZD mobile application group will be asked to download and use the W-GenZD mobile application that will provide information and tools through a chatbot (a computer program designed to communicate with users). Participants will be invited to use the mobile application as often as they like during the 4-week treatment period - we will encourage 5 to 10 minutes of daily use.
  W-GenZD Mobile Application: Woebot for Adolescents (W-GenZD) is a mobile application program that delivers evidence-based therapy for the symptoms of mild-moderate depression and anxiety in adolescents in brief "conversations" with a fully automated relational agent called Woebot. It is a brief, self-guided 4 week-intervention that draws from cognitive behavioral therapy (CBT), interpersonal psychotherapy for adolescents (IPT-A), and elements of dialectical behavior therapy (DBT), depending on the presenting situation, to help the adolescent develop emotion regulation skills in the context of their everyday life. In this way, the mobile application is designed to be targeted, relevant, and integrated into the lived experience of adolescents, capable of delivering the appropriate technique for the problem at hand, at the time of need.
Period: Overall Study
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group
Started | 71 | 70
Completed | 69 | 65
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- CBT-Lite Teletherapy Group: Participants assigned to the CBT-Lite teletherapy group will be asked to attend 1-hour teletherapy group sessions over Zoom once a week for 4 weeks. In this group, a study clinician will cover topics such as building a coping tool box, accepting your feelings, challenging negative thoughts, and problem solving.
  CBT-Lite Teletherapy: The CBT-Lite teletherapy group is a brief, 4-week intervention held once weekly for an hour, and limited to those triaged into the Children's Hospital of the King's Daughters low-intensity track and participating in this protocol. An assigned study clinician will facilitate each teletherapy group with approximately 10 adolescents in each session. Each group begins with orientation and reviewing group rules, individual check-ins with each participant (rating stress level and hopefulness), followed by a guided mindfulness moment. Sessions are designed to draw from elements of cognitive behavioral therapy (CBT) and the 4 topics include: building a coping tool box, accepting your feelings, challenging negative thoughts, and problem solving.
- Total: Total of all reporting groups
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group | Total
Number analyzed (Participants) | 71 | 70 | 141
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 13 years | 14 | 14 | 28
  Age, Categorical: 14 years | 25 | 19 | 44
  Age, Categorical: 15 years | 17 | 14 | 31
  Age, Categorical: 16 years | 9 | 19 | 28
  Age, Categorical: 17 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 54 | 110
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 24 | 24 | 48
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Hispanic | 9 | 2 | 11
  Mixed Race | 4 | 2 | 6
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Other | 1 | 0 | 1
  White | 29 | 40 | 69
Gender Identity [Count of Participants; unit: Participants]
  Agender | 0 | 2 | 2
  Different identity | 1 | 2 | 3
  Genderqueer | 1 | 0 | 1
  Man/boy | 22 | 17 | 39
  Non-binary | 1 | 4 | 5
  Prefer not to answer | 2 | 3 | 5
  Woman/girl | 44 | 42 | 86
Sexual Orientation [Count of Participants; unit: Participants]
  Asexual | 2 | 0 | 2
  Bisexual | 9 | 11 | 20
  Don't know | 5 | 1 | 6
  Lesbian or gay | 2 | 5 | 7
  Pansexual | 8 | 5 | 13
  Pansexual; Asexual | 2 | 0 | 2
  Prefer not to answer | 2 | 2 | 4
  Queer | 1 | 1 | 2
  Straight or heterosexual | 40 | 45 | 85
Highest Education Level [Count of Participants; unit: Participants]
  Elementary or middle school (grades 1-8) | 26 | 24 | 50
  High school graduate or GED (grade 12) | 1 | 3 | 4
  Some high school (grades 9-11) | 44 | 43 | 87
Primary Presenting Problem at Intake [Count of Participants; unit: Participants]
  Anxiety | 37 | 39 | 76
  Depression | 34 | 31 | 65
Concomitant Medications [Count of Participants; unit: Participants]
  Currently Taking Antidepressants | 10 | 11 | 21
  Currently Taking Antipsychotics | 0 | 0 | 0
  Currently Taking Stimulants | 8 | 8 | 16
Caregiver Relationship to Participant [Count of Participants; unit: Participants]
  Legal guardian | 3 | 5 | 8
  Parent | 68 | 65 | 133
Caregiver Employment Status [Count of Participants; unit: Participants]
  Employed, full time | 41 | 44 | 85
  Employed, part time | 8 | 4 | 12
  Not employed, looking for work | 4 | 2 | 6
  Not employed, not looking for work | 0 | 3 | 3
  On disability, not able to work | 2 | 2 | 4
  Prefer not to answer | 4 | 4 | 8
  Primary care-taker at home, not employed outside of the home | 11 | 8 | 19
  Retired | 1 | 3 | 4
Caregiver Marital Status [Count of Participants; unit: Participants]
  Divorced / Separated | 18 | 11 | 29
  Married / Partnered / Cohabiting | 36 | 43 | 79
  Prefer not to answer | 0 | 4 | 4
  Single | 14 | 11 | 25
  Widowed | 3 | 1 | 4
Caregiver Insurance Type [Count of Participants; unit: Participants]
  Medicaid and similar insurance | 26 | 13 | 39
  Medicare | 1 | 2 | 3
  Multiple sources | 4 | 3 | 7
  No insurance | 1 | 0 | 1
  Prefer not to answer | 0 | 2 | 2
  Private insurance | 30 | 36 | 66
  TRICARE or other military health care | 6 | 14 | 20
  VA: Past and present | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Usage Rating Profile-Intervention Revised (URP-IR), Feasibility Subscale
Description: Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Items (e.g., "The total time required to do the treatment procedures was manageable") are rated on a 6-point Likert scale (1 = "strongly disagree" to 6 = "strongly agree"). Total feasibility scores range from 6-36, with higher scores indicating greater intervention feasibility with the W-GenZD mobile application or the CBT-Lite teletherapy groups.
Time Frame: End-of-treatment (4 weeks from baseline)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group
Number analyzed (Participants) | 71 | 70
score on a scale | 30.00 [28.50 to 31.50] | 30.00 [28.20 to 31.80]

2. Primary Outcome: Usage Rating Profile-Intervention Revised (URP-IR), Acceptability Subscale
Description: Measure of acceptability. A 9-item subscale that inquires about intervention acceptability. For the purposes of this study, an adapted 6-item version of the subscale was utilized. Items (e.g., "This treatment is an effective choice for addressing a variety of depression concerns) are rated on a 6-point Likert scale (1 = "strongly disagree" to 6 = "strongly agree"). Total acceptability scores range from 6-36, with higher scores indicating greater intervention acceptability with the W-GenZD mobile application or the CBT-Lite teletherapy groups.
Time Frame: End-of-treatment (4 weeks from baseline)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group
Number analyzed (Participants) | 71 | 70
score on a scale | 28.00 [26.05 to 29.95] | 29.10 [26.70 to 31.51]

3. Secondary Outcome: Patient Health Questionnaire, 8 Items (PHQ-8)
Description: Measure of depression severity. An 8-item abbreviated version of the PHQ-9 used to assess depressive symptomatology over the past 2 weeks. The PHQ-8 excludes an item assessing suicidality. Items (e.g., "Over the last 2 weeks, how often have you been bothered by ... feeling down, depressed or hopeless?") are rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day"). Total scores range from 0-24, with higher scores indicating increased severity of depressive symptoms.
Time Frame: Baseline; end-of-treatment (4 weeks from baseline); change from baseline to end-of-treatment at 4 weeks
Population: Multiple imputation used for missing scores at end-of-treatment at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- W-GenZD Mobile Application Group: Participants assigned to the W-GenZD mobile application group will be asked to download and use the W-GenZD mobile application that will provide information and tools through a chatbot (a computer program designed to communicate with users). Participants will be invited to use the mobile application as often as they like during the 4-week treatment period - we will encourage 5 to 10 minutes of daily use.
  W-GenZD Mobile Application: W-GenZD is a mobile application program that delivers evidence-based therapy for the symptoms of mild-moderate depression and anxiety in adolescents in brief "conversations" with a fully automated relational agent called Woebot. It is a brief, self-guided 4 week-intervention that draws from cognitive behavioral therapy (CBT), interpersonal psychotherapy for adolescents (IPT-A), and elements of dialectical behavior therapy (DBT), depending on the presenting situation, to help the adolescent develop emotion regulation skills in the context of their everyday life. In this way, the mobile application is designed to be targeted, relevant, and integrated into the lived experience of adolescents, capable of delivering the appropriate technique for the problem at hand, at the time of need.
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group
Number analyzed (Participants) | 71 | 70
score on a scale
  PHQ-8 at Baseline | 10.65 (6.31) | 11.16 (5.20)
  PHQ-8 at Week 4 (EOT) | 8.75 (4.91) | 9.42 (4.88)
  PHQ-8 Change from Baseline to Week 4 (EOT) | -1.89 (4.83) | -1.74 (4.33)
Statistical Analysis 1: Comparison: W-GenZD Mobile Application Group vs CBT-Lite Teletherapy Group; Test type: Non-Inferiority — The non-inferiority (NI) test for the secondary outcome (i.e., PHQ-8 Week 4 EOT score) was assessed using the pre-specified NI margin of 2.0. NI of W-GenZD to CBT-Lite was declared if the upper bound of the one-sided 97.5% confidence interval (CI) was less than 2; Mean Difference (Net) = -0.67, 95% CI 2-sided [-2.30 to 0.96]

ADVERSE EVENTS:
Time Frame: Throughout study (from baseline through 8 weeks)
Description: Safety was monitored via: 1) concerning language detection within each intervention; 2) biweekly phone check-ins by the research coordinator with the caregiver; 3) spontaneous report to study personnel. Upon learning of a potential safety concern, on-call licensed study personnel contacted the caregiver to assess the adolescent's safety, identify the level of intervention needed, and provide resources as needed. Participants were withdrawn if they were deemed to require a higher level of care.
Arm/Group | W-GenZD Mobile Application Group | CBT-Lite Teletherapy Group
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/70
Other Adverse Events (participants affected / at risk) | 2/71 | 2/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | W-GenZD Mobile Application Group (N=71) | CBT-Lite Teletherapy Group (N=70)
Adverse Event, Mild Severity (Psychiatric disorders) | 1 (1) | 1 (1)
Adverse Event, Moderate Severity (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT05372913/Prot_SAP_000.pdf